CLINICAL TRIAL: NCT04744480
Title: Effect of Topical Anesthesia Combined With Intravenous Induction on Hemodynamics During the Induction Period in Patients Undergo Cardiac Surgery: a Randomized Controlled Study
Brief Title: Effect of Topical Anesthesia on Hemodynamics During the Induction Period in Patients Undergo Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TACTICS
Record Dates: First submitted 2021-01-24; First posted 2021-02-09 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease; Arrhythmia; Myocardial Disease
Keywords: Topical anesthesia; Cardiac surgery; Hemodynamics; Induction period
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Arrhythmias, Cardiac; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combined topical anesthesia induction group (Experimental): The superior glottic mucosa would be anesthetized 3 times with a vaporizer before intravenous anesthesia. After the intravenous induction, a catheter would be inserted to provide the subglottic anesthesia，3-5ml 2% lidocaine would be used for supraglottic anesthesia, and 3ml 1% tetracaine would be used for subglottic anesthesia.
  Interventions: Procedure: The combined topical anesthesia induction group
- The routine induction group (No Intervention): The superior glottic mucosa would be anesthetized 3 times with a vaporizer before intravenous anesthesia. After the intravenous induction, a catheter would be inserted to provide the subglottic anesthesia.In the routine induction group，all procedures will be the same as those of the topical anesthesia group, The drug will be replaced with constant volume saline.

INTERVENTIONS:
Procedure: The combined topical anesthesia induction group — The superior glottic mucosa would be anesthetized 3 times with a vaporizer before intravenous anesthesia. After the intravenous induction, a catheter would be inserted to provide the subglottic anesthesia，3-5ml 2% lidocaine would be used for supraglottic anesthesia, and 3ml 1% tetracaine would be used for subglottic anesthesia.
  Arms: The combined topical anesthesia induction group

SUMMARY:
The aim of the induction is to decrease stress response of endotracheal intubation. It is also important to keep hemodynamics stable during and after the induction period. Previous studies have shown that topical anesthesia can provide excellent superior supraglottic and subglottic local anesthetic effects and can significantly reduce the dosage of intravenous anesthetics. Therefore, it is significant to explore whether the combination of topical anesthesia and intravenous anesthetics could decrease the stress response of endotracheal intubation and keep hemodynamics stable during and after the induction period.

DETAILED DESCRIPTION:
The routine anesthesia induction strategy for cardiac surgery is to decrease stress response during endotracheal intubation by using large doses of opioids. However, high doses of opioids often leads to persistent and recurrent hypotension in patients from the anesthesia induction period to the beginning of the surgery. Patients scheduled to accept cardiac surgery often have severe concomitant disease. Hemodynamic fluctuation might lead to disastrous events. Anesthesia induction for such patients should not only provide adequate depth of anesthesia to decrease the stress response of endotracheal intubation, but also make hemodynamics stable after tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to accept elective /major cardiac surgery;
2. Patients older than 18 years and younger than 85 years;
3. Patients of The American Society of Anesthesiologists ( ASA )Ⅱ - Ⅳ level grade;
4. Patients signed the informed consent form for the clinical study;

Exclusion Criteria:

1. Patients cannot cooperate to topical anesthesia;
2. Patients with a left cardiac assist device prior to surgery;
3. Patients with aortic dissection;
4. Patients with Intra Aortic Balloon Pump (IABP) prior to surgery;
5. Patients treated with Extracorporeal Membrane Oxygenation (ECMO) prior to surgery;
6. Patients with difficult airway;
7. Patients with high sensitivity and hypersensitivity to lidocaine and tetracaine;
8. Patients with atrioventricular block;
9. Hemoglobin(Hb)<80g/L；
10. Patients who have participated in other clinical studies during the last 3 months;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
The area under the curve of baseline blood pressure | From the beginning of general anesthesia induction(T1) to the surgery beginning(T2). T1 is when induction drug (midazolam) is administered. T2 is defined as the time of the skin incision. It will take up to 1hour or 2hours.
  The area under the curve (AUC) of blood pressure below baseline from the beginning of general anesthesia induction to the surgery beginning.

SECONDARY OUTCOMES:
The frequency and types of vasoactive drugs used. | From the beginning of general anesthesia induction(T1) to the surgery beginning(T2). T1 is when induction drug (midazolam) is administered. T2 is defined as the time of the skin incision. It will take up to 1hour or 2hours.
  The frequency and types of vasoactive drugs used ,such as the use of norepinephrine and dopamine.
The incidence of arrhythmias. | From the beginning of general anesthesia induction(T1) to the surgery beginning(T2). T1 is when induction drug (midazolam) is administered. T2 is defined as the time of the skin incision. It will take up to 1hour or 2hours.
  The incidence of arrhythmias, such as atrioventricular block, atrial fibrillation, ventricular tachycardia and so on.
cardiac systolic function:Left Ventricular Ejection Fraction (LVEF) | Preoperative, intraoperative
  Left ventricular ejection fraction is a reliable indicator of left ventricular systolic function. left ventricular ejection fraction (LVEF) (﹪)= stroke output (SV)/ left ventricular end-diastolic volume (LEDV)×100﹪
cardiac diastolic function:E/E' (the ratio of E peak and E') or E/A :(the ratio of E peak and A peak) | Preoperative, intraoperative
  E/A ratio, one of the main indicators for evaluating diastolic function, indicated normal diastolic function when E/A >1, and decreased diastolic function when E/A < 1.
cardiac output monitoring indicator: CO(cardiac output) | Intraoperative
  CO＝Stroke Output (SV)× Heart Rate (HR).The relevant parameters are obtained by the cardiac output monitor which produced by Edwards Lifesciences.
cardiac output monitoring indicator: SVV(stroke volume variation) | Intraoperative
  The relevant parameters are obtained by the cardiac output monitor which produced by Edwards Lifesciences.
cardiac output monitoring indicator: CI(cardiac index) | Intraoperative
  CI＝CO/ Body Surface Area (BSA).The relevant parameters are obtained by the cardiac output monitor which produced by Edwards Lifesciences.
cardiac output monitoring indicator: SVR (systemic vascular resistance) | Intraoperative
  SVR＝60×(MAP-CVP)/CO. MAP: mean arterial pressure. CVP: central venous pressure.The relevant parameters are obtained by the cardiac output monitor which produced by Edwards Lifesciences.
The number of patients with postoperative hoarseness. | Three days after the surgery
  Hoarseness was classified as mild, moderate and severe according to the severity.
The number of patients with postoperative sore throat. | Three days after the surgery
  Sore throats can be evaluated using the Numeric Pain Scale (NRS) pain numerical score.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lv, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Meng-Lv, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen TT, Lv M, Wang JH, Wei CS, Gu CP, Wang YL. Addition of topical airway anaesthesia to conventional induction techniques to reduce haemodynamic instability during the induction period in patients undergoing cardiac surgery: protocol for a randomised controlled study. BMJ Open. 2022 Jan 25;12(1):e053337. doi: 10.1136/bmjopen-2021-053337. PMID 35078841